CLINICAL TRIAL: NCT06615635
Title: A Pivotal, Single Arm, Open Label Clinical Study to Assess the Safety and Efficacy of Intratumoral Alpha DaRT224 for the Treatment of Immunocompromised Patients With Cutaneous Squamous Cell Carcinoma
Brief Title: Clinical Study Protocol for Cutaneous SCC for Immunocompromised Patients
Acronym: DaRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPT-SCC-04
Record Dates: First submitted 2024-09-22; First posted 2024-09-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Squamous Cell Carcinoma; Alpha Radiation; Immunocompromised; Carcinoma, Squamous; Skin Cancer; Brachytherapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an International Multicenter, Pivotal, Single Arm, Open Label pivotal trial with DaRT for the treatment of Immunocompromised Cutaneous Squamous Cell Carcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- DaRT seeds (Experimental): Diffusing Alpha emitters Radiation (DaRT) treatment to be delivered through radioactive sources inserted into malignant cutaneous squamous cell carcinoma of Immunocompromised Patients
  Interventions: Device: DaRT seeds

INTERVENTIONS:
Device: DaRT seeds — Diffusing Alpha emitters Radiation (DaRT) treatment to be delivered through radioactive sources inserted into malignant cutaneous squamous cell carcinoma of Immunocompromised Patients
  Other Names: DaRT

SUMMARY:
This is a multi-center clinical study enrolling up to 28 participants. The primary objectives are to determine the objective response rate (ORR) established by the confirmed best overall response (BOR) following intratumoral administration of DaRT - Diffusing Alpha-Emitters Radiation Therapy. Secondary objectives are to:

1. Determine Progression Free Survival (PFS) up to 12 months after Alpha DaRT sources insertion.
2. Assess Overall Survival (OS) of patients treated with DaRT up to 12 months.
3. Assess Local control up to 12 months after DaRT insertion.

DETAILED DESCRIPTION:
This study is a pivotal multicenter, single arm, open label clinical study to assess the efficacy and safety of intratumoral Alpha DaRT-224 for the treatment of of Immunocompromised Patients with Cutaneous Squamous Cell Carcinoma

The "Diffusing Alpha-emitter Radiation Therapy (DaRT)", based on the intratumoral placement of an encapsulated Radium-224 source (3.7 days half-life), is described in this study. These sources release short-lived alpha-emitting atoms into the tumor microenvironment by recoil. Alpha DaRT sources will be inserted into Cutaneous Squamous Cell Carcinoma tumors and will be removed following 14-21 days.

The The objective response rate (ORR), which is calculated as the percent of patients achieving an objective response. Best overall response using the Response Evaluation Criteria in Solid Tumors guidelines (RECIST v1.1). Best overall response is assessed starting from DaRT removal. Safety will be assessed based on the cumulative incidence rate, severity and outcome of device related Adverse Events (AEs). Classification of AEs will be done according to CTCAE v5.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with cutaneous SCC histologically confirmed 2. Histopathological confirmation within 6 months of enrollment provided no tumor treatment occurred between the biopsy and enrollment 3. Immunocompromised due to any primary or secondary immunodeficiencies Measurable disease according to RECIST v 1.1.

  4. Patient able and willing to undergo multiple CT scans 5. Tumor size ≤7 cm, at the longest diameter. 6. Single lesion per subject. 7. Targeted lesion must be technically amenable for complete coverage (including margins) by the DaRT seeds. Targets will be deemed technically amenable for complete coverage if there are entry and exit vectors for placement that are not hindered by bone or major vessels or other vital organs (eg. eye) as decided by treating physician and sponsor.

  8. Interstitial implant indication validated by multidisciplinary team. 9. ECOG Performance Status ≤2. 10. Life expectancy ≥12 months. 11. Subjects male/ female ≥18. 12. Willing and have the ability to provide signed Informed Consent. 13. Patients, male and female, with reproductive potential (including women who are menopausal for less than a year and not surgically sterilized), must practice acceptable effective methods of birth control, such as barrier methods, condom or diaphragm with spermicide or abstinence. Birth control should be continued for 1 year after the DaRT insertion visit.

  14. Women with childbearing potential must provide a negative pregnancy test during the screening period and up to V1, prior to the DaRT insertion procedure.

  15. Blood tests values:
  * Platelets ≥100,000 mm3,
  * Total bilirubin ≤ 1.5xULN,
  * AST ≤2.5xULN,
  * SGOT ≤2.5xULN,
  * SGPT ≤2.5xULN,
  * Alkaline Phosphatase ≤2.5xULN.
  * Creatinine Clearance ≥30 ml/min.
  * INR or Prothrombin time ≤1.5xULN.

Exclusion Criteria:

* 1. Distant or nodal metastatic disease (according to the TNM staging system - N+ or M1 patients are excluded).

  2. T4 disease 3. extensive PNI 4. Previously untreated cutaneous SCC 5. Mucosal SCC. 6. Inability to fully cover the entire volume with DaRT seeds 7. Inability to place DaRT seeds into tumor due to inaccessibility by presence of bones or major vessels or vital organs 8. Inability or unwillingness to undergo multiple CT scans 9. Patients receiving any of the following within 4 weeks of enrollment:
  1. Antineoplastic systemic chemotherapy or biological therapy
  2. Immunotherapy
  3. Investigational agents other than the study intervention
  4. Radiation therapy
  5. Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial.

     10. Longest tumor diameter >7 cm. 11. Tumor with keratoacanthoma histology. 12. Known hypersensitivity to any component of treatment. 13. Clinically significant cardiovascular disease e.g., cardiac failure of New York Heart Association class III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, history of myocardial infarction in the last 12 months.

     14. Any medical or Psychiatric illness, which in the opinion of the investigator would compromise the patient's ability to tolerate treatment and to adhere to the clinical trial protocol.

     15. Serious medical comorbidities that, in the opinion of the investigator, may affect subject compliance and/or interpretation of treatment safety or effectiveness.

     16. High probability of protocol non-compliance (in opinion of investigator). 17. Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.

     18. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.

     19. Patients do not agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry and for 1 year after the DaRT insertion visit.

     20. Breastfeeding or pregnant women 21. Tattoos scars, body jewelry (e.g., nose rings) or other identifying marks which cannot be adequately hidden on digital photos or other identifying marks which cannot be adequately hidden on digital photos

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate | From Day 14 until 52 weeks
  • Assessment of the objective response rate (ORR) determined by the best overall response using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1).

SECONDARY OUTCOMES:
Progression Free Survival | Up to 12 months after DaRT seed insertion
  • Determine Progression Free Survival (PFS) up to 12 months after DaRT seed insertion.
Overall Survival | Up to 12 months after DaRT seed insertion
  • Assess Overall Survival (OS) of patients treated with DaRT up to 12 months.
Local control | Up to 12 months after DaRT seed insertion
  • Assess Local control up to 12 months after DaRT insertion.

OTHER OUTCOMES:
Safety Objectives | Up to 12 months following DaRT insertion
  Assess the safety of the Alpha DaRT treatment, based on the cumulative incidence rate, severity and outcome of device related AEs. Classification of AEs will be done according to CTCAE v5.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Banner Health, Gilbert, Arizona
  - Us Dermatology Parthners, Phoenix, Arizona
  - Alliance Dermatology, Phoenix, Arizona
  - Integrity Research Clinical Associates, Boca Raton, Florida
  - Hollywood Dermatology, Hollywood, Florida
  - Palm Beach Dermatology Group, Palm Beach, Florida
  - Day Star Skin Cancer Center, Poinciana, Florida
  - Emory University, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Bassett Healthcare, Cooperstown, New York
- Hadassah Medical Center, Jerusalem, Israel